CLINICAL TRIAL: NCT03448055
Title: Nutritional Intervention With the Cysteine-rich Whey Protein Isolate Dietary Supplement Immunocal® in MCI Patients: Promotion of Brain Health & Wellness During Aging and Oxidative Stress
Brief Title: Nutritional Intervention With the Dietary Supplement, Immunocal® in MCI Patients: Promotion of Brain Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunotec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MCI-IMM15
Record Dates: First submitted 2018-02-06; First posted 2018-02-27 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: MCI, AD, MRI, GSH, Immunocal, brain health, neuropsychological evaluation
MeSH Terms: conditions — Cognitive Dysfunction; Glucocorticoid-Remediable Aldosteronism

STUDY DESIGN:
Intervention Model Description: Nutritional supplemetation with Immunocal 20gm daily for 6 months (180 days)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Other): Immunocal 20gm daily
  Interventions: Dietary Supplement: Immunocal

INTERVENTIONS:
Dietary Supplement: Immunocal — cysteine-rich whey protein isolate

SUMMARY:
Alzheimer disease (AD) is a dementing illness characterized by progressive neuronal degeneration, gliosis, and the accumulation of intracellular inclusions and extracellular deposits of amyloid in discrete regions of the basal forebrain, hippocampus, and the association cortices. Mild cognitive impairment (MCI) refers to individuals with cognitive impairment (often memory loss) that fails to meet clinical criteria for AD or another dementing illness.

ELIGIBILITY:
This study is recruiting Mild Cognitive Impaired (MCI) patients from the Memory Clinic of the Jewish General Hospital only.

Inclusion Criteria:

Subjects meeting diagnostic criteria for MCI:

* Age 55-85
* Male or female
* Non-smoker

To ensure that the subject can physically fit in the scanner:

1. body weight ≤ 120 kg and
2. with a linear dimension max 55cm (shoulders or belly) Expected to remain in the greater Montreal area for the duration of study.

Exclusion Criteria:

* Presence of an active, systemic illness (e.g., cancer, rheumatoid arthritis, etc.) or other chronic neurological (e.g. Parkinson's disease, multiple sclerosis) or psychiatric (e.g. major depression, schizophrenia) disease.
* Subjects taking other experimental medications or psychotropic agents.
* Subjects with MRI contraindications such as pacemaker, aneurysm clips, artificial heart valves, metal fragments, foreign objects or claustrophobia.
* Ambulatory subjects: As wheelchair-bound subjects present additional difficulties for transportation and MRI scanning.

Musculoskeletal abnormalities that preclude the ability of the subject to lie on his/her back for 1hr during MRI scanning.

* Subjects who have a protein restricted diet as per their medical history.
* Pregnancy
* Subjects using N-acetylcysteine, α-lipoic acid supplements, other whey protein supplements or Vitamin C, within 2 months of enrolment and during the entire 6 months study period.
* Allergies to milk proteins/ Milk protein intolerance

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2022-11-25 (Estimated); Study Completion 2023-11-25 (Estimated)

PRIMARY OUTCOMES:
Change in GSH levels in the brain | Baseline compared to month 6 (180 days)
  Change in cerebral Glutathione levels of MCI patients measured by MRI/MRS scans

SECONDARY OUTCOMES:
Change in plasma GSH:GSSG ratios measured by HPLC | Baseline compared to month 6 (180 days)
  To evaluate positive correlation between plasma GSH:GSSG ratios and changes in cerebral GSH
Evaluation of neuropsychological and cognitive functions | Baseline compared to month 6 (180 days)
  The Memory Clinic of JGH Neuropsychological evaluation questionnaire will be used to measure both neuropsychological and cognitive functions

CONTACTS AND LOCATIONS:
Locations (1):
- Memory Clinic/Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song W, Tavitian A, Cressatti M, Galindez C, Liberman A, Schipper HM. Cysteine-rich whey protein isolate (Immunocal(R)) ameliorates deficits in the GFAP.HMOX1 mouse model of schizophrenia. Free Radic Biol Med. 2017 Sep;110:162-175. doi: 10.1016/j.freeradbiomed.2017.05.025. Epub 2017 Jun 8. PMID 28603087
- [Background] Winter AN, Ross EK, Daliparthi V, Sumner WA, Kirchhof DM, Manning E, Wilkins HM, Linseman DA. A Cystine-Rich Whey Supplement (Immunocal(R)) Provides Neuroprotection from Diverse Oxidative Stress-Inducing Agents In Vitro by Preserving Cellular Glutathione. Oxid Med Cell Longev. 2017;2017:3103272. doi: 10.1155/2017/3103272. Epub 2017 Aug 15. PMID 28894506